CLINICAL TRIAL: NCT02521116
Title: Comparison of Retinal Oxygenation and Retinal Vessel Diameters in Healthy Subjects and Patients With Diabetic Retinopathy or Retinal Vein Occlusion Between DVA and Oxymap
Acronym: DVA-Oxymap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AUGEN-061014
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects; Diabetic Retinopathy; Retinal Vein Occlusion
Keywords: retinal oxygenation; retinal vessel diameters; Dynamic vessel analyzer (DVA); Oxymap T1
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Vein Occlusion

ARMS (1):
- Healthy subjects (Other): healthy study subjects, age 18-80 years
  Interventions: Other: Dynamic Vessel Analyzer; Other: Oxymap T1

INTERVENTIONS:
Other: Dynamic Vessel Analyzer
Other: Oxymap T1

SUMMARY:
To date two different instruments are commercially available to measure retinal oxygen saturation and retinal vessel diameters: Dynamic Vessel Analyzer (DVA) and Oxymap. Retinal oxygen saturation analysis is based on spectroscopic evaluation of retinal fundus images. Up to now no data comparing both instruments for the measurement of retinal oxygen saturation and vessel diameter are available in the literature.

Study objectives: To compare retinal oxygenation and retinal vessel diameters in healthy subjects and patients with diabetic retinopathy or retinal vein occlusion between 2 commercially available systems (DVA, Oxymap T1)

Study design: Open pilot study

Study population:

30 healthy volunteers, age 18-80 years 30 type 2 diabetic patients with mild or moderate non-proliferative diabetic retinopathy, age 18-80 years 30 patients with retinal vein occlusion, age 18-80 years

Topically administered medication:

Tropicamide (Mydriaticum "Agepha"®, Agepha, Vienna, Austria), dose: 1-2 drops per study day for dilation of the pupil Oxybuprocainhydrochloride combined with sodium fluorescein (Thilorbin®, Alcon Pharma GmbH, Freiburg, Germany), dose: 1 drop in one eye for measurements of intraocular pressure Nonylacidvanillylamide combined with Nicotinic-acid--ß-butoxyethylester (Finalgon®, Boehringer Ingelheim RCV GmbH & Co KG, Vienna, Austria): topical on the earlobe

Methods:

Dynamic vessel analyzer Oxymap T1 Blood pressure and pulse rate measurement Applanation tonometry Oxygen and carbon dioxide partial pressure measurement in arterialized blood from earlobe

Main outcome variables:

Difference of oxygen saturation of retinal vessels between DVA and Oxymap T1

The motive for this investigation is to compare data between 2 commercially available instruments for the measurement of retinal oxygen saturation and retinal vessel diameter in healthy subjects as well as in patients with ocular disease associated with altered retinal oxygenation. Comparative data from both systems are currently not available. Data from this study will allow the comparison of studies performed with different systems. All oxygen measurement procedures are non-invasive and painless. Hence, the risk/benefit ratio appears to be acceptable.

ELIGIBILITY:
Inclusion criteria healthy volunteers

* normal ophthalmic findings, ametropia < 3 dpt
* men and women aged between 18 and 80 years

Exclusion Criteria:

Any of the following will exclude a subject from the study:

* participation in a clinical trial in the 3 weeks preceding the study
* symptoms of a clinically relevant illness in the 3 weeks before the first study day
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01-03 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Difference of oxygen saturation of retinal vessels between DVA and Oxymap T1 | participants will be followed for the duration of outpatient clinic visit, an expected average of 1 days

SECONDARY OUTCOMES:
Difference of retinal vessel diameter between DVA and Oxymap T1 | participants will be followed for the duration of outpatient clinic visit, an expected average of 1 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria